CLINICAL TRIAL: NCT02917252
Title: Ketone Bodies Ingested Orally Alter Metabolism for Glucose, Lipid, and Protein
Brief Title: How Orally Consumed 3-hydroxybuturate Alters Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: RM-1-10-72-157-16
Record Dates: First submitted 2016-09-27; First posted 2016-09-28 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2016-09

CONDITIONS: Acute Ketosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Subjects drink 3-hydroxybuturate
  Interventions: Other: 3-hydroxybuturate
- Placebo (Placebo Comparator): Subjects drink saline
  Interventions: Other: Placebo

INTERVENTIONS:
Other: 3-hydroxybuturate — Drink of ketone bodies
  Arms: Intervention
Other: Placebo — Drink of saline
  Arms: Placebo

SUMMARY:
This study evaluate the metabolic effects of orally ingested ketone bodies. The study is conducted as a randomized, cross over study.

DETAILED DESCRIPTION:
Subject participate for two separate days; i) intervention, ii) placebo. Intervention: subjects drink ketone body solution. Tracer kinetics on glucose and lipid metabolism is applied. Muscle tissue and adipose tissue biopsies are taken.

Placebo: subjects drink saline. Same sampling as on intervention day.

ELIGIBILITY:
Inclusion Criteria:

* BMI 20-30

Exclusion Criteria:

* Smoking
* alcohol or drug abuse
* Critically ill

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-04-03 (Actual); Study Completion 2017-04-03 (Actual)

PRIMARY OUTCOMES:
3-hydroxybuturate | 0-270 minutes
  blood level of 3-hydroxybuturate

SECONDARY OUTCOMES:
Glucose | 0-270 minutes
  Glucose tracer kinetics, endogenous glucose production, muscle biopsy
lipid metabolism | 0-270 minutes
  Palmitate tracer kinetics, free fatty acid accumulation, adipose tissue biopsies

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Svart M, Rittig N, Pedersen SB, Jessen N, Moller N. Oral 3-hydroxybutyrate ingestion decreases endogenous glucose production, lipolysis, and hormone-sensitive lipase phosphorylation in adipose tissue in men: a human randomized, controlled, crossover trial. Diabet Med. 2021 Feb;38(2):e14385. doi: 10.1111/dme.14385. Epub 2020 Sep 22. PMID 32794582